CLINICAL TRIAL: NCT00846989
Title: A 4-week Multi-center, Single-masked, Randomized, Latanoprost-controlled, Parallel Group Study to Assess the Efficacy, Tolerability and Safety of RKI983 (0.05% and 0.10%) Ophthalmic Solution Given Twice a Day Versus Once Daily Latanoprost 0.005%, in Patients With Primary Open Angle Glaucoma or Ocular Hypertension.
Brief Title: Efficacy, Tolerability and Safety of RKI983 (0.05% & 0.10%) vs Xalatan in Patients With POAG or Ocular Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRKI983A2201
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2013-02

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: glaucoma,; primary open-angle glaucoma (POAG),; ocular hypertension (OH),; intraocular pressure (IOP)
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Glaucoma, Open-Angle | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: RKI983A
- 2 (Experimental)
  Interventions: Drug: RKI983A
- 3 (Active Comparator)
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: RKI983A — RKI983 0.05 % twice daily
  Arms: 1
Drug: RKI983A — RKI983 0.1 % twice daily
  Arms: 2
Drug: Latanoprost — Latanoprost 0.005 % once a day
  Arms: 3

SUMMARY:
This purpose of this study is to access the efficacy, tolerability and safety of RKI983 (0.05% and 0.10%) ophthalmic solution bid versus once daily latanoprost 0.005%, in patients with POAG or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Females must be post-menopausal or surgically sterile, or must use concomitantly two acceptable forms of effective contraception
* Clinical diagnosis of POAG or OH
* For study eyes not previously treated with anti-glaucoma medications

  * IOP must be ≥ 22 mm Hg at least at two assessment time-points at Screening, and
  * IOP must be ≥ 22 mm Hg at least at two assessment time-points at Baseline, and
  * IOP must be ≥ 20 mm Hg and ≤ 36 mm Hg at all Screening and Baseline assessment time-points.
* Or for study eyes previously treated with anti-glaucoma medications

  * IOP must be ≥ 14 mm Hg and ≤ 24 mm Hg at least at two assessment time-points at Screening.
  * IOP must be ≥ 22 mm Hg at least at two assessment time-points at Baseline (after wash-out)
  * IOP must be ≥ 20 mm Hg and ≤ 36 mm Hg at all Baseline assessment time-points

Exclusion Criteria:

* History of or current clinically significant ocular conditions in either eye that would contraindicate the use of an investigational drug or latanoprost (e.g. active intraocular inflammation), or that might affect interpretation of the results of the study.
* History or presence of clinically significant medical problems that contraindicate the use of an investigational drug or latanoprost, including but not limited to:

  * Uncontrolled hypertension with systolic blood pressure ≥ 160 mm Hg and/or diastolic blood pressure ≥ 100 mm Hg measured at more than one blood pressure reading at Screening or Baseline;
  * myocardial infarction within the 3 months period prior to randomization;
  * active severe viral infections such as active encephalitis, meningitis, hepatitis, herpes simplex, or herpes zoster (minor viral upper respiratory infections such as colds do not require exclusion.)
* Presence of moderate or severe (grade 2 or 3) conjunctival hyperemia in the study eye at Baseline Visit.
* Argon laser trabeculoplasty or any prior IOP lowering surgery in the study eye.
* Ocular surgery in the study eye within 3 months prior to the Screening Visit.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Mean reduction of the daily average intraocular pressure (IOP) . | from Baseline to Day 29

SECONDARY OUTCOMES:
Mean IOP reduction at each assessment time-point | from Baseline to Day 8, 15, 22 and 29
Mean reduction of the daily average IOP | from Baseline to Days 8, 15 and 22
Frequency of adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- United States (28):
  - Novartis Investigative Site, Artesia, California
  - Novartis Investigative Site, Inglewood, California
  - Novartis Investigative Site, La Jolla, California
  - Novartis Investigative Site, Poway, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Danbury, Connecticut
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Morrow, Georgia
  - Novartis Investigative Site, Roswell, Georgia
  - Novartis Investigative Site, Kaneohe, Hawaii
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Bossier City, Louisiana
  - Novartis Investigative Site, Cambridge, Massachusetts
  - Novartis Investigative Site, Springfield, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Bethpage, New York
  - Novartis Investigative Site, Lynbrook, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Mt. Pleasant, South Carolina
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, El Paso, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Spokane, Washington

REFERENCES:
- See also: Results for CRKI983A2201 can be found on the Novartis Clinical Trial Results website. — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2938